CLINICAL TRIAL: NCT01720888
Title: A Controlled Open Label Phase II Study Assessing the Efficacy of Intracoronary Autologous Mesenchymal Stem Cells in Patients With Ischemic Dilated Cardiomyopathy
Brief Title: Intracoronary Autologous Mesenchymal Stem Cells Implantation in Patients With Ischemic Dilated Cardiomyopathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National University of Malaysia (Other)
Collaborators: Cytopeutics Sdn. Bhd. (Industry)
Responsible Party: Principal Investigator, Professor Dr Oteh Maskon, Professor, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERGS/1/2011/SKK/UKM/02/72
Record Dates: First submitted 2012-11-01; First posted 2012-11-02 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Ischemic Dilated Cardiomyopathy
Keywords: Autologous; Bone Marrow; Mesenchymal Stem Cells; Ischemic Dilated Cardiomyopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Maximal medical therapy (No Intervention): Maximal medical therapy which comprises of optimal pharmacological therapy
- Maximal medical therapy and BM-MSCs (Experimental): Autologous Bone marrrow-derived mesenchymal stem cells implantation
  Interventions: Other: BM-MSCs

INTERVENTIONS:
Other: BM-MSCs — Intracoronary implantation of bone marrow-derived mesencymal stem cells
  Other Names: Bone marrow-derived mesenchymal stem cells implantation
  Arms: Maximal medical therapy and BM-MSCs

SUMMARY:
Despite the recent advances in medical and surgical treatment, heart failure resulting from ischemic cardiomyopathy (ICM) remains the leading cause of cardiovascular mortality. Ischemic dilated cardiomyopathy(ICM) is defined as abnormally enlarged left ventricular (LV) cavity with documented poor LV function as a result of severe coronary artery disease (CAD). LV remodelling which is inevitable after an infarct has been postulated to contribute largely to the poor outcome of patients with ICM, therefore prevention of LV remodelling is the goal for the treatment in patients with severe CAD. Cell therapy represents a novel therapeutic strategy for treating cardiac diseases including severe CAD and heart failure. A type of stem cells known as mesenchymal stem cells(MSCs)can be isolated from bone marrow.This study aims to test the differentiation potential and therapeutic capacity of MSC from severe CAD patients after intracoronary implantation in an ischemic myocardial environment in Malaysian population.

DETAILED DESCRIPTION:
Ischemic dilated cardiomyopathy(ICM) is defined as abnormally enlarged left ventricular (LV) cavity with documented poor LV function as a result of severe coronary artery disease (CAD). LV remodelling which is inevitable after an infarct has been postulated to contribute largely to the poor outcome of patients with ICM, therefore prevention of LV remodelling is the goal for the treatment in patients with severe CAD. Cell therapy represents a novel therapeutic strategy for treating cardiac diseases including severe CAD and heart failure. A type of stem cells known as mesenchymal stem cells(MSCs)can be isolated from bone marrow. Experimental and clinical studies to date have shown that mesenchymal stem cells represent the most suitable cell type for regeneration therapy after myocardial infarction (MI). After injection into ischemic myocardium, bone marrow-derived MSC (BM-MSC) from various animal species can differentiate into multiple cell lineages, including endothelial cells and cardiomyocytes, thereby improving LV function.

In Malaysia we have previously demonstrated our capability in isolating and extracting MSC from a small volume of bone marrow aspirates.The isolation, expansion and feasibility of storage, transport and differentiation of human MSC for clinical application has been performed locally. The researchers used autologous BM-MSC, ex vivo expanded, on three patients with end-stage ischemic dilated cardiomyopathy who were on the heart transplant waiting list and each patient was injected with MSCs directly into the myocardium during open heart surgery. After twelve months, all patients remained alive and well with significant improvement in cardiac function, quality of life and other parameters including reduction of myocardial scar volume as seen from cardiac scans.

The same group of researchers further carried out a study on ten patients with severe dilated cardiomyopathy and refractory cardiac function despite maximum medical therapy to receive autologous BM-MSC implantation via intramyocardial or intracoronary route. All patients remained alive at 1 year while recorded significant improvements in LV ejection fraction and other LV parameters from baseline to 6 and 12 months. Reduction in scar was also noted in six of the patients by 12 months.

Following these results, this study aims to test the differentiation potential and therapeutic capacity of MSC from severe CAD patients after intracoronary implantation in an ischemic myocardial environment in Malaysian population.

ELIGIBILITY:
Inclusion Criteria:

* aged between 35 to 75 years
* diagnosed to have ICM confirmed by previous coronary angiogram showing significant coronary artery disease >70% or history of previous myocardial infarction.
* myocardial infarction event occured 6 months or longer from time of screening.
* LV ejection fraction of ≤40% by echocardiogram or cardiac MRI.

Exclusion Criteria:

* Likelihood of heart failure from other causes such as idiopathic, infective or metabolic cardiomyopathy,valvular heart disease and pericardial disease.
* patients who had undergone a coronary artery bypass graft(CABG) procedure.
* patients who do not have any visible/significant myocardial scar.
* patients with any cardiovascular metallic implantation.
* any contraindication to bone marrow aspiration
* any contraindication to coronary contrast angiography and angioplasty.
* any acute or chronic communicable diseases including Hepatitis B, Hepatitis C and HIV.
* any past history of neoplasia and primary haematological disease.
* any current, past or paroxysmal cardiac arrhythmias.
* renal impairment indicated by creatinine clearance of less than 30 ml/min.
* liver impairment indicated by serum alanine transferase level at 4 times greater than normal value.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Change in LV ejection fraction as measured by echocardiogram and cardiac MRI after implantation | 1 month, 3 months, 6 months, 9 months, 12 months

SECONDARY OUTCOMES:
Changes in functional status | 12 months
Improvement in other LV parameters as assessed by echocardiogram and cardiovascular magnetic resonance(CMR). | 1 months, 3 months, 6 months, 9 months, 12 months
Resolution of scar tissue volume/area on cardiac MRI | 6 months, 12 months.
Change in serum N Terminal-pro B type natriuretic peptide(NT-proBNP)level | 1 month, 6 months, 12 months
Freedom from major adverse cardiac events as defined by myocardial infarction, hospitalization for angina, myocardial infarction or heart failure, or death (all cause of mortality). | 1 month, 3 months, 6 months, 9 months, 12 months

OTHER OUTCOMES:
No peri-procedural complications | 1 month, 3 months, 6 months, 9 months, 12 months
Significant improvement in overall left ventricular function | 12 months
Resolution of scar tissue | 6 months, 12 months
Reduction of major adverse cardiac events | 1 month, 3 months, 6 months, 9 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Oteh Maskon, MB Bch, Principal Investigator — Universiti Kebangsaan Malaysia Medical Centre
Locations (1):
- UKM Medical Centre, Cheras, Kuala Lumpur, Malaysia